CLINICAL TRIAL: NCT02374502
Title: Increasing Physical Activity in Ankylosing Spondylitis (INPACT-AS): a Randomised Controlled Trial
Brief Title: Increasing Physical Activity in Ankylosing Spondylitis: a Randomised Controlled Trial
Acronym: INPACT-AS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Tom O'Dwyer, Lead Investigator, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC2015/01/02
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Spondylitis, Ankylosing
Keywords: Spondylarthropathies; Motor Activity; Physical Therapists; Accelerometry
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthropathies; Motor Activity | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Intervention Group (Experimental): Participants in this intervention group will receive a twelve week 'Brief Intervention' delivered by a physiotherapist. Participants will have an initial consultation with a physiotherapist, followed by a number of follow-up sessions. The number and timing of follow-up sessions will be at the participant's discretion (a minimum of 3 and a maximum of 11 over the duration of the study). The follow-up sessions can be face-to-face, over the telephone, or video conferencing depending on participant preference. Participants may additionally opt-in for a weekly email or text message reminder of physical activity goals.
  Interventions: Behavioral: Brief Intervention
- Control Group (No Intervention): Participants in this control group will be asked to continue with their current levels of physical activity.

INTERVENTIONS:
Behavioral: Brief Intervention — 'Brief Intervention' is the term used to mean verbal advice, discussion, negotiation or encouragement, with or without written or other support or follow-up. 'Brief Interventions' provide a structured way to deliver advice and involve the provision of formal help and follow-up. They aim to equip people with tools to change attitudes and handle underlying problems.
  Arms: Brief Intervention Group

SUMMARY:
Ankylosing spondylitis is a chronic inflammatory condition that mostly affects the spine. This results in back pain and stiffness, and causes difficulty with daily activities. Physical activity and exercise are key components of the management of ankylosing spondylitis, however many adults with ankylosing spondylitis do not meet physical activity recommendations. This study aims to investigate the effects of a twelve week intervention designed to increase physical activity and exercise in adults with ankylosing spondylitis.

DETAILED DESCRIPTION:
Participants will be randomly allocated to one of two groups. An intervention group will receive individual consultations with a physiotherapist. The aim of the meetings will be to motivate and support participants on an individual basis, with the goal of increasing weekly physical activity. The second group, the control group, will continue with their current management strategies. All participants will be assessed at baseline, post-intervention (after twelve weeks) and after a three month follow-up period. The primary outcome measure will be free-living physical activity over one week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis (diagnosed by a rheumatologist).
* Able to read and understand the English language.
* On stable pharmacological management.

Exclusion Criteria:

* Under 18 years of age, or over 64 years of age
* Unable to read and understand the English language
* Concomitant cardiac, respiratory or neurological condition
* Co-morbidity restricting physical activity or inability to ambulate without a mobility aid
* Acute lower limb injury
* Uncontrolled epilepsy
* Cognitive difficulties limiting ability to follow safety and protocol instructions
* Pregnant
* Change in medication (type of dosage) within six weeks of testing
* On beta-blocker medication.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Free-living Physical Activity | up to 12 weeks follow-up
  Actigraph monitor GT3X-BT worn during waking hours over 7 days.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | up to 12 weeks follow-up
Bath Ankylosing Spondylitis Functional Index (BASFI) | up to 12 weeks follow-up
Bath Ankylosing Spondylitis Global score (BAS-G) | up to 12 weeks follow-up
Ankylosing Spondylitis Quality of Life questionnaire (ASQoL) | up to 12 weeks follow-up
Cardiorespiratory capacity | up to 12 weeks follow-up
  VO2peak measured by submaximal, incremental treadmill test
Body Composition | up to 12 weeks follow-up
  Bioelectric impedance analysis & waist/hip circumference
Flexibility | up to 12 weeks follow-up
  Bath Ankylosing Spondylitis Metrology Index (BASMI) & Chest Expansion
Muscular fitness | up to 12 weeks follow-up
  Push-up test and curl-up test
Exercise Barriers and Beliefs Scale (EBBS) | up to 12 weeks follow-up
Arthritis self-efficacy questionnaire (Ankylosing Spondylitis version) | up to 12 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Finbar O'Shea, Principal Investigator — St. James's Hospital, Ireland; Fiona Wilson, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Trinity Centre for Health Sciences, Dublin, Ireland

REFERENCES:
- [Derived] O'Dwyer T, Monaghan A, Moran J, O'Shea F, Wilson F. Behaviour change intervention increases physical activity, spinal mobility and quality of life in adults with ankylosing spondylitis: a randomised trial. J Physiother. 2017 Jan;63(1):30-39. doi: 10.1016/j.jphys.2016.11.009. Epub 2016 Dec 8. PMID 27989730